CLINICAL TRIAL: NCT01373567
Title: An Open Label, Non-comparative, Multicentre, Phase IV Study to Evaluate the Safety, Tolerability and Efficacy of Tinefcon in Patients With Plaque Psoriasis
Brief Title: A Phase IV Clinical Trial to Study the Safety, Tolerability and Efficacy of Tinefcon in Patients With Plaque Psoriasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Piramal Enterprises Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TINEFCON/49/10
Record Dates: First submitted 2010-12-07; First posted 2011-06-15 (Estimated); Last update posted 2012-11-22 (Estimated); Status verified 2012-11

CONDITIONS: Plaque Psoriasis
Keywords: Plaque Psoriasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TINEFCON (Experimental): Tablets of 700 mg.
  Interventions: Drug: TINEFCON

INTERVENTIONS:
Drug: TINEFCON — Two 700 mg tablets of Tinefcon in the morning and evening to be taken orally.

SUMMARY:
Psoriasis is a chronic inflammatory hyperproliferative disease of the skin affecting approximately 2% of the world's population.This phase IV study is planned to monitor performance of Tinefcon in patients suffering from psoriasis under conditions of actual use and fulfill requirements to monitor all adverse drug reactions (ADRs) in psoriasis patients treated with Tinefcon. This study will add to literature on the risks and benefits of Tinefcon the novel oral TNF-alpha release inhibitor.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of at least 18 years of age with clinical diagnosis of plaque psoriasis
* Subject who understand and willing to sign informed consent document before start of any study specific assessment

Exclusion Criteria:

* Pregnant and lactating females
* Subject with active infection, acute or chronic due to bacteria, viruses, fungi or parasites (most notably tuberculosis, and chronic hepatitis B)
* Subject with heart failure (New York Heart Association class III or IV)
* Subject with demyelinating disease
* Subject with solid cancer or hematologic malignancy diagnosed within last 5 years with a potential for progression
* Women of childbearing potential [defined as a sexually mature woman who has not undergone hysterectomy or who has not been naturally postmenopausal for at least 24 consecutive months (i.e. who has had menses any time in the preceding 24 consecutive months)] and men, not agreeing to use adequate contraception (e.g., hormonal or barrier method of birth control or abstinence) after signing an informed consent document (ICD), during the duration of study participation and for at least 4 week after withdrawal from the study, unless they are surgically sterilized
* Subject with situations associated with a high risk of infection such as latent untreated tuberculosis, joint prosthesis infection within last 12 months, indwelling urinary catheter, uncontrolled diabetes, chronic obstructive pulmonary disease, skin ulcer
* Subject with known premalignant lesions (such as polyps in the colon or urinary bladder, cervical dysplasia and myelodysplasia)
* Subject known to be seropositive and/or clinically suspected to have the human immunodeficiency virus infection
* Subject with any condition that might make it difficult for the subject to participate in the study, at the discretion of the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 298 (Actual)
Dates: Start 2010-12; Primary Completion 2012-02 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Change in Psoriasis area severity index score | At week 4, week 8 and week 12 or early termination
  Change from baseline at week 4, week 8 and week 12 or early termination

SECONDARY OUTCOMES:
Gene expression profiling and Immunohistochemistry | At baseline and week 12 or early termination
Physicians global assessment score | At week 4, week 8 and week 12 / early termination visit
Nail psoriasis severity index | At baseline and at week 12 or early termination
Psoritic arthritis evaluation | At baseline and week 12 or early termination

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Sharmila Patil, Principal Investigator — D.Y.Patil Medical college and Hospital, Dept. of Dermatology & STD,Sector-5, Nerul, Navi Mumbai; Dr. Jerajani, Principal Investigator — Lokmanya Tilak Municipal Medical College & General Hospital, Department of Dermatology, First Floor, College Building,Sion, Mumbai-400022 India; Dr. Saple, Principal Investigator — Dr. Saple's clinic, 88, 3rd Lane, Hindu Colony, Near Bhagini Samaj, Dadar (East), Mumbai-400014; Dr.Ranjan Rawal, Principal Investigator — Sheth VS General Hospital, Department of Dermatology, Ellis Bridge, Ahmedabad -380006, Gujrat, India; Dr Sudhakar Grandhi, Principal Investigator — Medipoint Hospitals Pvt. Ltd.,Pentagon Research Pvt. Ltd, 241/1, New DP Road, Aundh, Pune-411007, Maharashtra; Dr Sushil Pande, Principal Investigator — NKP Salve Institute and Lata Mangeshkar Hospital,Nagpur; Dr. Torsekar, Principal Investigator — Rajiv Gandhi Medical College & CSMH,Department of Dermatology, Kalwa, Thane; Dr. C.R. Srinivas, Principal Investigator — PSG Hospital,Department of Skin & STD,Avinashi Road, Peelamedu, Coimbatore, Tamilnadu-641004; Dr. DVS Pratap, Principal Investigator — Durgabai Deshmukh Hospital & Research Center, Andhramahila Sabha Road, Vidyanagar, University Road,Hyderabad; Dr. Aruna Samarth, Principal Investigator — Sai Skin Care Clinic, H.No.:2-1-409, Nallakunta, O.U.Road, Hyderabad; Dr. Kanwar, Principal Investigator — Postgraduate Institute of Medical Education and Research,Department of Dermatology ,Venerology & Leprology,Sector-12-Chandigarh; Dr. Meetesh Agarwal, Principal Investigator — 178/DH Sector, Scheme No. 74, Vijaynagar, Indore 452 2010; Dr. Kailash Bhatia, Principal Investigator — Bhatia Skin Center,124-128, Anand Bazar, Bima Nagar, Indore; Dr. Parmjit Singh Walia, Principal Investigator — DR WALIA'S SKIN & LASER CLINIC, SCF - 30, PHASE; Dr. Bhavesh Swarnkar, Principal Investigator — Swarnkar Superspeciality Centre,84,Shreenagar Main,Regency Avenue,Ground Floor, Near Anand Bazar,Indore; Dr. Sandesh Gupta, Principal Investigator — Skin & Laser Center,F-12/10 Krishna Nagar, New Delhi; Dr. Puneet Goyal, Principal Investigator — Renova Skin & Laser Clinic,Sector 9, Shopping Centre,Opposite Meera Marg, Madhyam Marg, Mansarovar, Jaipur; Dr.Rizwan Haq, Principal Investigator — Radiance Skin Care Clinic, Opp. Muslim Library,Tekdi Road, Sadar, Nagpur; Dr Vikrant Saoji, Principal Investigator — Navprabhat Chambers,Opp. Tarun Bharat,Central Bazar Road,Ramdaspeth, Nagpur; Dr.B. Leelavathy, Principal Investigator — M.S. Diabetes and Shirdi Skin care centre 6/1, 80 Feet Road, Opp. Krishna Sagar Hotel, Indiranagar, Bangalore; Dr Titarmare, Principal Investigator — Skin Care Clinic, Consultant Dermatologist &Venerologist,Akshay Towers(Basement), Umrer Road,Sakkardhara Square, Nagpur; Dr Shatrughan Sahay, Principal Investigator — Sri Skin Care & Laser Clinic,Netaji Subash Chandra Bose Complex, Tulsidas Marg (Opp. Charak Pathalogy) Chowk-Lucknow
Locations (23):
- India (23):
  - Durgabai Deshmukh Hospital & Research Center, Hyderabad, Andhra Pradesh
  - Postgraduate Institute of Medical Education and Research,Department of Dermatology ,Venerology & Leprology, Chandigarh, Chandigarh
  - Sheth VS General Hospital, Department of Dermatology, Ahmedabad, Gujarat
  - M.S. Diabetes and Shirdi Skin care centre, Bangalore, Karnataka
  - Bhatia Skin Center,124-128, Anand Bazar, Bima Nagar, Indore, Madhtya Pradesh
  - Scheme No. 74, , Vijaynagar, ,, Indore, Madhya Pradesh
  - Swarnkar Superspeciality Centre,84,Shreenagar Main,Regency Avenue,Ground Floor, Near Anand Bazar, Indore, Madhya Pradesh
  - Sai Skin Care Clinic, Hyderabad, Maharashtra
  - Dr. Saple's clinic, Mumbai, Maharashtra
  - Lokmanya Tilak Municipal Medical College & General Hospital, Department of Dermatology, First Floor, College Building,Sion, Mumbai, Maharashtra
  - Seth GS Medical College &KEM Hospital,Department of Dermatology, Mumbai, Maharashtra
  - Dr.Vikrant Saoji,27, Navprabhat Chambers,Opp. Tarun Bharat,Central Bazar Road,Ramdaspeth, Nagpur, Maharashtra
  - NKP Salve Institute and Lata Mangeshkar Hospital, Nagpur, Maharashtra
  - Radiance Skin Care Clinic, Nagpur, Maharashtra
  - Skin Care Clinic, Consultant Dermatologist &Venerologist, Nagpur, Maharashtra
  - Medipoint Hospitals Pvt. Ltd, Pune, Maharashtra
  - Rajiv Gandhi Medical College, Thane, Maharashtra
  - Skin & Laser Center,F-12/10 Krishna Nagar,, New Delhi, New Delhi
  - Dr Walia'S Skin & Laser Clinic, Scf - 30, Phase- 3B-2, S.A.S. Nagar, Mohali, Punjab
  - Renova Skin & Laser Clinic,Sector 9, Shopping Centre,Opposite Meera Marg, Madhyam Marg, Jaipur, Rajasthan
  - PSG Hospital,Department of Skin & STD, Coimbatore, Tamil Nadu
  - Sri Skin Care & Laser Clinic, Lucknow, Uttar Pradesh
  - D.Y.Patil Medical college and Hospital, Dept. of Dermatology & STD,Sector-5, Nerul, Navi Mumbai